CLINICAL TRIAL: NCT01033591
Title: Rationale and Design of a Randomised Controlled Trial Evaluating the Effectiveness of an Exercise Program to Improve the Quality of Life of Patients With Heart Failure in Primary Care: The EFICAR Study Protocol
Brief Title: Exercise for Patients With Heart Failure in Primary Care: the EFICAR
Acronym: EFICAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Basque Health Service (Other Government)
Collaborators: Carlos III Health Institute (Other Government); Preventive Services and Health Promotion Research Network (Other); Castilla-La Mancha Health Service (Other); Castilla-León Health Service (Other); Public Health Service of Cataluña (Other); Islas Baleares Health Service. (Unknown)
Responsible Party: Principal Investigator, Jesus Torcal Laguna, general practitioner, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFICAR PS09/01498 -RD06/0018
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Heart Failure
Keywords: Primary Health Care; Family PractiCe; Hearth Failure; Exercise; Randomized Controlled Trials; Multicenter Study; Quality of life
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Supervised exercise + Optimized treatment according to the European Society of Cardiology guidelines
  Interventions: Behavioral: Supervised progressive exercise program with an aerobic and a strength component + Optimized treatment
- Control (Other): Optimized treatment according to the European Society of Cardiology guidelines
  Interventions: Behavioral: Optimized treatment according to the European Society of Cardiology guidelines

INTERVENTIONS:
Behavioral: Supervised progressive exercise program with an aerobic and a strength component + Optimized treatment — Three month supervised progressive exercise program with an aerobic (high intensity intervals) and a strength component; and the programme will continue linked with community resources for 9 months
  Arms: Exercise
Behavioral: Optimized treatment according to the European Society of Cardiology guidelines — Optimized treatment according to the European Society of Cardiology guidelines
  Arms: Control

SUMMARY:
Quality of life decreases as the heart failure worsens and is one of the biggest worries of these patients. Physical exercise has been shown as a safe intervention for people with heart failure. Previous studies have tested heterogeneous exercise programs using different QoL instruments and reported that the effects on QoL are inconsistent. The aim of this study is to evaluate the effectiveness of a new exercise program for people with heart failure (EFICAR), additional to the recommended optimal treatment in primary care, to improve QoL, functional capacity and cardiovascular risk factor control.

DETAILED DESCRIPTION:
Multicenter clinical trial in which 150 patients with heart failure in NYHA class II-IV will be randomized to two parallel groups: EFICAR and control. After being recruited, through the reference cardiology services, in six health centres from the Spanish Primary Care Prevention and Health Promotion Research Network (redIAPP), patients are followed for 1 year after the beginning of the intervention. Both groups receive the optimized treatment according to the European Society of Cardiology guidelines. In addition, the EFICAR group performs a 3 month supervised progressive exercise program with an aerobic (high-intensity intervals) and a strength component; and the programme continues linked with community resources for 9 months. The main outcome measure is the change in health-related QoL measured by the SF-36 and the Minnesota Living with Heart Failure Questionnaires at baseline, 3, 6 and 12 months. Secondary outcomes considered are changes in functional capacity measured by the 6-Minute Walking Test, cardiac structure (B-type natriuretic peptides), muscle strength and body composition. Both groups will be compared on an intention to treat basis, using multi-level longitudinal mixed models. Sex, age, social class, co-morbidity and cardiovascular risk factors will be considered as potential confounding and predictor variables.

Protocol for the intervention group The EFICAR group differs from the control group only in terms of the exercise programme, which has two phases. The exercise programme is a combination of "high-intensity interval training" and "muscular strength training". It has been demonstrated that high intensity aerobic exercise leads to better aerobic and cardiovascular changes than light/moderate exercise in patients with HF • 1st PHASE (12 weeks, 3 sessions/week): for the first three months, patients carry out a progressive exercise programme of 36 sessions under the supervision of the nurse, starting at low intensity (first month) and increasing it month by month.

Aerobic training: Aerobic exercise is undertaken on a cycloergometer, including warm-up, conditioning and cool down phase. From the beginning, the exercise sessions are personalised according to the physical condition of each patient. The first month is for "start-up", the second for "progress" and the third for "maintenance". For those patients that are very weak or are not used to aerobic exercise, the first sessions are of light-to-moderate intensity.

The Borg scale is used to evaluate the "perception of effort" during and after each session (values ranging between 6 and 20). This is a very useful scale to determine intensity with beta blockers, auricular fibrillation, pace-makers or other conditions which may alter the normal response of the heart rate to exercise. The exercise is also monitored with respect to the emergence of symptoms. Aerobic exercise is done before the strength training to guarantee activation of the muscles and cardiovascular system.

Muscular strength training: muscular strength work is a essential aspect of the rehabilitation of patients with HF. To avoid training-related increase of the hemodynamic load the exercise is isotonic. In each session, after 5 min of stretching and 8-12 min of aerobic exercise, six types of exercise are carried out to work various muscle groups: biceps, upper arms and shoulders, knee extensors and flexors, hip flexors and extensors, and plantar flexors. For muscular strength training, weights are used for upper body and resistance bands for the lower body. A different percentage of body weight is applied for each muscular group. Each patient is regularly informed of the progress they have made.

• 2nd PHASE: The training given in the first phase is intended to ensure that the patients make this exercise part of their routine. They are trained to carry out a type of interval aerobic exercise to they can keep up in their own environment, indefinitely and independently, together with muscular strength exercises. In addition, they are taught how to self-regulate the exercise intensity (Borg Scale, pulsometers, symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤85 years.
* Diagnosis of HF on the basis of signs and symptoms (Framingham criteria) and evidence of structural heart alterations detected by echocardiography (Echo). Echo scanning guarantees that we are dealing with patients suffering from HF avoiding confounding clinical factors.
* Left ventricle ejection fraction < 50%.
* NYHA functional class II-IV, or Stages C of the American Heart Association, in a stable situation for at least the previous four weeks, with no changes in baseline functional status, no signs of congestion or changes in weight faster than 2 kg in three days.
* Receiving optimal treatment with angiotensin converting enzyme inhibitors (ACEI), angiotensin II receptor antagonists (ARA-II), beta blockers, diuretics, and aldosterone antagonists at stable doses for the previous four weeks, as long as there are no justified contraindications for their use, and meeting the clinical practice guidelines of the European Society of Cardiology.
* Anticoagulated patients without atrial fibrillation, ejection fraction < 30%, presence of intracardiac thrombi, or history of embolism.
* In cases of sinusal rhythm or atrial fibrillation, ventricular response is under control both at rest and during exercise (90 beats/minute at rest, and 130 beats/minute during moderate exercise).
* Absence of arrhythmia in exercise stress test that would contraindicate exercise.
* Obtain at least 4 METS at Naughton exercise test
* Able to attend an exercise programme and travel to the reference laboratory.
* Informed consent confirmed in writing.

Exclusion Criteria:

* Physical and mental comorbidity which prevents undertaking the exercise programme.
* Major cardiovascular events (in the previous 6 weeks) or cardiovascular procedures, including cardiac resynchronization or implantation of a defibrillator.
* Heart failure pending intervention (mitral valve replacement/repair, ventricular reconstruction, pacemaker/ resynchronization pacemaker, implantable defibrillator, transplant), given that the procedures greatly change the baseline functional status and the prognosis of the disease.
* Heart failure secondary to congenital heart disease or hypertrophic obstructive cardiomyopathy, given that there is a formal contraindication for exercise in such clinical situations.
* Carrier of a fixed-rate pacemaker.
* Exercise test that contraindicates exercise for safety reasons, especially in the case of exercise-induced arrhythmia.
* Poor cognitive state, depression or psychiatric disorder that prevent adherence to an exercise programme.
* Inability to travelling to the health centre by their own means.
* Current or planned pregnancy in the next year
* Aortic stenosis or severe valve disease
* Perform an exercise equivalent to the proposed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life ( SF36 and 'Minnesota Living with Heart Failure Questionnaire') | One year follow up
  The HRQL questionnaire is measured blindly with self-administered questionnaires: the Spanish version of the SF-36 and MLHFQ. Both questionnaires will be filled out before and after the intervention. SF-36 generates an 8-dimension health profile and two summary scores for the physical and mental components. The 21 items from the MLHFQ record the perception of the patient in relation to how the HF affects the emotional, social, physical and mental dimensions of their HRQL. Both questionnaires have been validated in the Spanish population.

SECONDARY OUTCOMES:
Change in functional capacity (6 Minute Walking Test) | One year follow up
  The Test of the 6-minute applies to assess functional capacity, as well as a predictor of morbidity and mortality in people with moderate to severe HF. Most of the daily activities that the patients with IC are performed at submaximal exercise intensity, similar to this test is performed. In addition, as a method of controlling the intensity, this test is recommended using a Borg scale between "relatively easy" and "slightly hard"
Cardiac structural changes (B-type natriuretic peptide) | One year follow up
  Cardiac structural changes (levels of natriuretic peptide predictor)
Muscle strength (dynamometer) | One year follow-up
  Muscle strength was measured with a handgrip dynamometer adjustable (TKK-5001) in four measurements: baseline, at the end of the exercise program, at 6 and 12 months. The hand grip dynamometry is an objective method for measuring muscle strength and an indicator of the functional integrity of the upper extremity that correlates with overall body strength
Body composition (fat and muscular weight) | One year follow up
  Body Mass Index (BMI): Diagnoses and classifies obesity. Also called Quetelet index, is calculated with the values of the weight in kg and height in meters. BMI = weight / (height)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Torcal, Dr., Principal Investigator — Basauri Health Center. Basque Health Service
Locations (1):
- Primary Care Research Unit of Bizkaia (Basque Health Service), Bilbao, Bizkaia, Spain

REFERENCES:
- [Derived] Zuazagoitia A, Grandes G, Torcal J, Lekuona I, Echevarria P, Gomez MA, Domingo M, de la Torre MM, Ramirez JI, Montoya I, Oyanguren J, Pinilla RO; EFICAR Group (Ejercicio Fisico en la Insuficiencia Cardiaca). Rationale and design of a randomised controlled trial evaluating the effectiveness of an exercise program to improve the quality of life of patients with heart failure in primary care: The EFICAR study protocol. BMC Public Health. 2010 Jan 25;10:33. doi: 10.1186/1471-2458-10-33. PMID 20100317